CLINICAL TRIAL: NCT07402187
Title: The Effect of Productivity Training on Perceived Job Stress and Productivity Attitudes Among Nurses: A Randomized Controlled Experimental Study
Brief Title: "Productivity Training and Job Stress Among Nurses"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/16
Record Dates: First submitted 2025-12-12; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Occupational Stress; Productivity
Keywords: Nursing; job stress; Productivity; Randomized Controlled Trial
MeSH Terms: conditions — Occupational Stress | interventions — Nurses

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group design with pre-, post-, and follow-up assessments to evaluate the effects of a three-week productivity training program on nurses' perceived job stress and productivity attitudes.
Masking Description: This study is open-label. Due to the nature of the intervention (productivity training), neither participants nor researchers were blinded to group allocation. Both the experimental and control groups were aware of their group assignments. Data collection and analysis were conducted objectively according to the predefined proto.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Productivity Training Program (Experimental): Participants in the experimental group will receive a structured productivity training program lasting three weeks and totaling 20 hours. The training covers topics such as the concept of productivity in nursing, time and stress management, process improvement, teamwork, leadership, the use of digital tools, and coping with job stress. Each week, various teaching methods including lectures, case analyses, simulations, practical exercises, group work, and brainstorming sessions will be used. The program aims to enhance participants' cognitive, affective, and practical competencies related to productivity and stress management in nursing practice.
  Interventions: Behavioral: Productivity Training Program for Nurses
- No Training Control Group (No Intervention): Participants in the control group will not receive any training during the study period. They will complete the same pre-test, post-test, and follow-up assessments as the experimental group. After the completion of data collection, the productivity training materials will be made available to control group participants to ensure ethical fairness.

INTERVENTIONS:
Behavioral: Productivity Training Program for Nurses — The intervention consists of a structured productivity training program designed for nurses, delivered over three weeks (total 20 hours). The program includes interactive theoretical and practical sessions covering topics such as:
  The concept and scope of productivity in nursing, Time and stress management, Process improvement and teamwork, Leadership and performance support mechanisms, Coping with job stress and building psychological resilience, Use of digital tools and technology to enhance efficiency. Various teaching methods are employed, including lectures, simulations, case analyses, group discussions, applied exercises, and brainstorming. The program aims to improve nurses' cognitive, affective, and practical skills related to productivity, while reducing perceived job stress.
  Arms: Productivity Training Program

SUMMARY:
This study aims to examine the effect of productivity training on nurses' perceived job stress and attitudes toward productivity. It was designed as a randomized controlled experimental study with a pre-test, post-test, and follow-up design. The experimental group will receive a three-week structured productivity training program, while the control group will not receive any intervention during the same period. Data will be collected using the Personal Information Form, the Nurses' Attitudes Toward Productivity Scale, and the Perceived Job Stress Scale. It is hypothesized that nurses who participate in the productivity training will report lower perceived job stress and higher productivity attitudes compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse
* Being over 18 years old
* Working in the institution for at least 3 months
* Volunteering to participate in the study

Exclusion Criteria:

* Not being a nurse
* Being over 65 years old
* Not volunteering to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Nurses' Attitude Scale Regarding Productivity | Time Frame: At baseline (before the training), immediately after the 3-week productivity training program, and 3 months after the training.
  Nurses' attitudes toward productivity will be assessed using the Nurses' Attitudes Toward Productivity Scale (NAPTS), developed and validated by Göktepe and Baykal (2012).
  The scale consists of 39 items and five subscales: professional commitment, working conditions, job demands, teamwork, and rewarding.
  Items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  Total and subscale scores are converted to a 0-100 scale, with higher scores indicating a more positive attitude toward productivity, and lower scores indicating a negative attitude toward productivity.
  Minimum score: 0 Maximum score: 100

SECONDARY OUTCOMES:
Perceived Work Stress Scale (PWSS) | Time Frame: At baseline (before the training), immediately after the 3-week productivity training program, and 3 months
  Perceived job stress levels of the participants will be assessed using the Perceived Job Stress Scale (PJSS), originally developed by Cohen and Williamson (1988) and adapted into Turkish by Baltaş (1998).
  The scale consists of 15 items rated on a 5-point Likert scale. The total score is calculated by taking the mean score of the 15 items.
  Based on the mean score, stress levels are categorized into six groups:
  A (3.5-4.0) B (1.0-1.3) C (1.4-1.9) D (2.0-2.5) E (2.6-3.1) F (3.2-3.4) Higher scores indicate higher perceived job stress. Stress levels classified as A, B, E, and F are considered stress levels that may negatively affect work efficiency and threaten health, whereas C represents stress levels suitable for individuals who prefer low challenge, and D represents the optimal stress level for health and productivity.
  Minimum score: 1.0 Maximum score: 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çerçi, Dr. Öğretim Üyesi, Principal Investigator — bağlantısız
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Arel University, Istanbul, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive personal and occupational information about nurses. Data will be analyzed and reported in aggregate form only. Access to anonymized data may be considered upon reasonable request and ethics committee approval.

DOCUMENTS (2):
  • Study Protocol (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT07402187/Prot_000.pdf
  • Informed Consent Form (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT07402187/ICF_001.pdf